CLINICAL TRIAL: NCT03675230
Title: Study of Tomotherapy HD in Medulloblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XH-18-012
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-07

CONDITIONS: Medulloblastoma
Keywords: TOMO irradiation
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3DCRT (Active Comparator): This arm will be planned by 3DCRT to the treatment of the Medulloblastoma
  Interventions: Device: 3DCRT
- Tomotherapy HD，TOMO (Experimental): This arm will be planned by TOMO to the treatment of the Medulloblastoma
  Interventions: Device: Tomotherapy HD

INTERVENTIONS:
Device: Tomotherapy HD — Patients with Medulloblastoma receiving Tomotherapy
  Arms: Tomotherapy HD，TOMO
Device: 3DCRT — Patients with Medulloblastoma receiving Three-Dimensional Conformal Radiation Therapy
  Arms: 3DCRT

SUMMARY:
The aim of the study was to improve local control and long-term survival in children with medulloblastoma, reduce the side effects of treatment and improve quality of life.

DETAILED DESCRIPTION:
The technical advantages of Tomotherapy HD in the radiotherapy of children medulloblastoma (advantages in clinical operation and physics) were transformed into clinical advantages, and the possible mechanisms were explored.

ELIGIBILITY:
Inclusion Criteria:

* The patient was diagnosed as myeloblastoma by surgical pathology with definite pathological classification. MRI of the head and spinal cord before and after operation, with definite staging; Radiotherapy was performed within 28 days after surgery.

Exclusion Criteria:

* Previous radiotherapy in the whole brain, whole spinal cord or primary focus; Postoperative radiotherapy for more than 28 days.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
QoL(quality of life) | 2 years
  Changes in quality of life were assessed by EORTC QLQ-C30

SECONDARY OUTCOMES:
PFS (progression free survival) | 2 years
  from the first day of therapy to the date of disease progression or death from any cause, whichever was first (according the criterion of RECIST 1.1 ).
OS (overall survival) | 2 years
  from the first day of therapy to death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: mawei jiang, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- The Department of Radiation Oncology, Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No